CLINICAL TRIAL: NCT03219138
Title: Development of an Algorithm Using Clinical Tests to Avoid Post-operative Residual Neuromuscular Block
Brief Title: Algorithm of Muscle Function Tests to Detect Residual Neuromuscular Blockade.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: Technical University of Munich (Other); University Hospital Muenster (Other); University Hospital Schleswig-Holstein (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Christoph Unterbuchner, Principal Investigator, University of Regensburg
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: N° 1783/ 07
Record Dates: First submitted 2017-07-08; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Residual Curarization
Keywords: muscle function tests
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Intervention Model Description: During anaesthesia calibrated neuromuscular function is monitored using evoked EMG of the adductor pollicis muscle (immobilised forearm) with a NMT module by a non-blinded investigator. During surgery, the (blinded) attending anaesthesiologist administers maintenance doses of atracurium according to clinical needs, i.e. without knowing the TOFR.
  After surgery patients' trachea is extubated according to clinical judgement. Immediately after extubation blinded anaesthesiologist tests the patient. The postoperative evaluation of neuromuscular function consists of eight clinical tests applied in a random order.
  Thereafter, an uncalibrated acceleromyography (50 mA, 2 Hz) is started on the contralateral arm and TOF ratio is measured.
  During the validation part of the developed algorithm the anaesthesiologist additionally had to judge tactile fading of the adductor pollicis.
  If a patient had any clinical signs of neuromuscular dysfunction, reversal with neostigmine is administered.
Who Masked: Care Provider
Masking Description: Immediately after extubation the blinded anaesthesiologist (care provider), who performs anesthesia, tests the patient in the operating room.
  The blinded anaesthesiologist is unable to see the data on the EMG monitor and the movement of the adductor pollicis muscle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromyography (No Intervention): Neuromuscular function was monitored, using evoked electromyography of the adductor pollicis muscle with a neuromuscular transmission module by a non-blinded investigator.
- Acceleromyography (Experimental): Immediately after extubation the blinded anaesthesiologist tested with an uncalibrated acceleromyography on the contralateral arm.
  Interventions: Device: Acceleromyography

INTERVENTIONS:
Device: Acceleromyography — Use of an uncalibrated acceleromyography
  Arms: Acceleromyography

SUMMARY:
Objective neuromuscular monitoring is the gold standard to detect postoperative residual curarization (PORC). Many anesthesiologist just use qualitative neuromuscular monitoring or unreliable, clinical tests. Goal of this study is to develop an algorithm of muscle function tests to identify PORC

DETAILED DESCRIPTION:
Background: Quantitative neuromuscular monitoring is the gold standard to detect postoperative residual curarization (PORC). Many anesthesiologists, however, use insensitive, qualitative neuromuscular monitoring or unreliable, clinical tests. Goal of this multicentre, prospective, double-blinded, assessor controlled study is to develop an algorithm of muscle function tests to identify PORC.

Methods: After extubation a blinded anesthetist performs eight clinical tests in 165 patients. Test results are correlated to calibrated electromyography train-of-four (TOF) ratio and to a postoperatively applied uncalibrated acceleromyography. A classification and regression tree (CART) is calculated developing the algorithm to identify PORC. This is validated against uncalibrated acceleromyography and tactile judgement of TOF fading in separate 100 patients.

ELIGIBILITY:
Inclusion Criteria: The patients were scheduled for elective low risk surgical procedures:

* laparoscopic abdominal procedures
* orthopedic
* minor visceral surgery

Exclusion Criteria:

* participation in another study
* body mass index over 30
* history of neuromuscular diseases
* gastro-esophageal reflux disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2008-01-08 (Actual); Primary Completion 2009-07-25 (Actual); Study Completion 2009-07-25 (Actual)

PRIMARY OUTCOMES:
Clinical muscle function tests | Muscle function tests are performed immediately after extubation.
  Measurement of postoperative residual curarisation with clinical muscle function test:
  * time able to open the eyes
  * appearence of diplopic images
  * time able to stick out the tongue
  * spatula pressure test
  * time able to lift the head
  * time able to lift the arm
  * strength of the patient pressing the investigator's hand
  * ability to swallow 20 ml of water

SECONDARY OUTCOMES:
Uncalibrated acceleromyography | Uncalibrated acceleromyography is measured immediately after extubation.
  Contralateral to the electromyography arm an uncalibrated acceleremyography measures objectively postoperative residual curarisation by examination of the train of four ratio.
Qualitative neuromuscular measurement | Qualitative acceleromyography is measured immediately after extubation.
  Contralateral to the electromyography arm qualitative tactile judgement of the train of four stimulation was measured by acceleremyography to scale postoperative residual curarisation.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - 6Klinik für Anästhesiologie und Operative Intensivmedizin, Universitätsklinikum Schleswig-Holstein, Campus Kiel,, Kiel
  - Klinik für Anaesthesiologie, Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinik und Poliklinik für Anästhesiologie und operative Intensivmedizin, Universitätsklinikum Münster, Münster
  - Klinik für Anaesthesiologie und operative Intensivmedizin, Klinikum am Steinenberg, Steinenbergstr. 31, 72764 Reutlingen, Germany, Reutlingen
  - Klinik und Poliklinik für Anästhesiologie und Intensivtherapie, Universität Rostock, Rostock

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baillard C, Clec'h C, Catineau J, Salhi F, Gehan G, Cupa M, Samama CM. Postoperative residual neuromuscular block: a survey of management. Br J Anaesth. 2005 Nov;95(5):622-6. doi: 10.1093/bja/aei240. Epub 2005 Sep 23. PMID 16183681
- [Background] Baillard C, Bourdiau S, Le Toumelin P, Ait Kaci F, Riou B, Cupa M, Samama CM. Assessing residual neuromuscular blockade using acceleromyography can be deceptive in postoperative awake patients. Anesth Analg. 2004 Mar;98(3):854-7, table of contents. doi: 10.1213/01.ane.0000100150.84698.8c. PMID 14980952
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Kotake Y, Ochiai R, Suzuki T, Ogawa S, Takagi S, Ozaki M, Nakatsuka I, Takeda J. Reversal with sugammadex in the absence of monitoring did not preclude residual neuromuscular block. Anesth Analg. 2013 Aug;117(2):345-51. doi: 10.1213/ANE.0b013e3182999672. Epub 2013 Jun 11. PMID 23757472
- [Derived] Unterbuchner C, Blobner M, Puhringer F, Janda M, Bischoff S, Bein B, Schmidt A, Ulm K, Pithamitsis V, Fink H. Development of an algorithm using clinical tests to avoid post-operative residual neuromuscular block. BMC Anesthesiol. 2017 Aug 4;17(1):101. doi: 10.1186/s12871-017-0393-4. PMID 28778151